CLINICAL TRIAL: NCT06812130
Title: Surviving the Pediatric Intensive Care Unit (PICU): Long-term Study to Understand and Improve Outcomes of PICU Survivors and Their Families
Brief Title: Surviving the Pediatric Intensive Care Unit (PICU)
Status: Recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National University Hospital, Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Jan Hau Lee, Associate Professor, KK Women's and Children's Hospital
Other Study IDs: ECOS Ref: 2024-3978
Record Dates: First submitted 2025-01-16; First posted 2025-02-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Post Intensive Care Syndrome (PICS)
Keywords: PICS-p; Prospective Observational Cohort Study; Post Intensive Care Syndrome in Paediatrics (PICS-p)
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HOPE Cohort (PICU Survivors): Helping to Optimize Patients' Experiences (HOPE) after Pediatric Critical Illness Cohort Study [Sample Size: 240 participants]
  Interventions: Other: This is a non-interventional study.
- SHACK-S Cohort (Siblings of PICU Survivors): Singapore Health outcomes After Critical illness in Kids - Siblings (SHACK-S): Experiences and Health Outcomes of Siblings in the first 6 months after PICU discharge of a critically ill child. [Sample Size (Quantitative): 164 participants; Sample Size (Qualitative): 20 participants]
  Interventions: Other: This is a non-interventional study.

INTERVENTIONS:
Other: This is a non-interventional study. — This is a non-interventional study.

SUMMARY:
Improvement in pediatric intensive care unit (PICU) supportive care has led to improvement in clinical outcomes and decreased mortality in pediatric critical illness. However, PICU survivors are at risk of long-term health sequalae. Given the increased recognition of physical, cognitive, and psychological sequelae in PICU survivors, the concept of post-intensive care syndrome-pediatrics (PICS-p) has been proposed. Besides the PICU patient/survivor, the PICS-p framework also highlights the impacts of a child's critical illness has on the family. The impact of a PICU admission extends beyond the patient and parents, potentially affecting healthy siblings who are navigating their own developmental challenges. Healthy siblings may face emotional distress, increased responsibilities, and disruptions in their daily routines, all of which can contribute to long-term negative outcomes if unaddressed. Thus, this study consists of two cohorts to understand the long-term physical, cognitive, and psychological outcomes in PICU survivors and their families, and the short-term impacts on siblings of critically ill children.

DETAILED DESCRIPTION:
The objectives of Helping to Optimize Patients' Experiences (HOPE) after Pediatric Critical Illness Cohort Study are:

1. [Primary] To characterize physical and cognitive health outcomes of PICU survivors.
2. [Primary] To investigate subgroups of critically ill children who have poor medium-term physical and cognitive health outcomes.
3. [Primary] To elucidate risk factors for poor physical and cognitive health outcomes in PICU survivors.
4. [Exploratory] To investigate the impact of physical and cognitive health of PICU survivors on overall family health.

The objectives of Singapore Health outcomes After Critical illness in Kids - Siblings (SHACK-S): Health Outcomes and Experiences of Healthy Siblings in the first 6 months after PICU discharge are:

1. [Primary] To describe and compare quality-of-life in healthy siblings at 1, 3 and 6 months after PICU discharge.
2. [Primary] To explore the experiences and support needs of healthy siblings 6 months after PICU discharge of a critically ill child.
3. [Secondary] To examine the experiences of recovery trajectory of healthy siblings.

Thus, HOPE cohort will provide information and insight regarding which groups of PICU patients and associated PICU therapies are associated with the highest risk for poor survivorship. The conduct of this study will also allow us to identify the challenges and find appropriate solutions in performing a cohort study with an emphasis on patient-reported outcomes (e.g., functional status, cognition and quality of life). Concurrently, the SHACK-S cohort will provide insights to understand the impacts of PICU admission on siblings and their recovery.

ELIGIBILITY:
Inclusion Criteria:

[HOPE Cohort]

1. Between 28 days - 16 years of age at PICU admission
2. Have an expected PICU stay > 48 hours

[SHACK-S Cohort]

1. Healthy children (aged 4 -16 years old) with critically ill sibling between 28 days - 16 years of age at PICU admission
2. Has a critically ill sibling who has an expected PICU stay > 48 hours
3. Lives in the same household as the critically ill sibling and parents prior to admission

Exclusion Criteria:

[HOPE Cohort]

1. Do-Not-Resuscitate status
2. Lack of informed consent
3. Prior enrolment in this study

[SHACK-S Cohort]

1. Children of critically ill sibling with Do-Not-Resuscitate status
2. Children with condition listed on paediatric Complex Chronic Conditions (CCC) system Version 3.0 or with neurocognitive/neurodevelopmental delays or disorders
3. Previous admission to PICU
4. Lack of informed consent
5. Prior enrolment in this study

Ages: 28 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: [HOPE Cohort] Paediatric patients, aged 28 days - 16 years of age, admitted to either PICU at KK Women's and Children's Hospital, Singapore or National University Hospital, Singapore.
  [SHACK-S Cohort] Siblings, aged 4 - 16 years old, of paediatric patients admitted to either PICU at KK Women's and Children's Hospital, Singapore or National University Hospital, Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 404 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
[HOPE] Pediatric Evaluation of Disability Inventory (PEDI-CAT) [Physical health outcomes of PICU survivors] | Baseline, Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measures functional domains: Daily Activities, Mobility, Social/Cognitive and Responsibility
[HOPE] Functional Status Scale (FSS) [Physical health outcomes of PICU survivors] | Baseline, Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measures 6 domains of functioning: Mental Status, Sensory, Communication, Motor Function, Feeding, Respiratory
[HOPE] Hand-grip strength test [Physical health outcomes of PICU survivors] | Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measures of maximum voluntary muscle strength (Only for study participants aged 6 years old and above)
[HOPE] 6-minute walk test [Physical health outcomes of PICU survivors] | Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Assessment of aerobic capacity and endurance (Only for study participants aged 6 years old and above)
[HOPE] Developmental Profile-4 (DP-4) [Cognitive outcomes of PICU survivors] | Baseline, 6-, 12- and 18-month post-PICU discharge
  Measures developmental domains: Physical, Adaptive Behaviour, Social-Emotional, Cognitive and Communiation
[HOPE] Bayley Scales of Infant and Toddler Development - 4th edition (Bayley-4) [Cognitive outcomes of PICU survivors] | 6- and 18-month post-PICU discharge
  Measures developmental domains: Cognitive and Language (Only for study participants aged below 3 years old)
[HOPE] National Institute of Health Toolbox - Cognition Battery (NIHTB-CB) [Cognitive outcomes of PICU survivors] | Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measures cognitive health (Only for study participants aged 3 years old and above)
[HOPE] Strengths and Difficulty Questionnaire (SDQ) [Cognitive outcomes of PICU survivors] | Baseline, 6-, 12- and 18-month post-PICU discharge
  Screening tool for behavioural and emotional problems (Only for study participants aged 2 years old and above)
[SHACK-S] PedsQL 4.0 Short Form 15 (SF5) [Quality of Life in Siblings of Critically Ill Children] | PICU discharge, 1-, 3-, and 6-month post-PICU discharge
  Measures generic health-related quality of life in children
[SHACK-S] Strengths and Difficulties Questionnaire (SDQ) [Experiences and Support Needs of Siblings of Critically Ill Children] | 1-, 3-, and 6-month post-PICU discharge
  Screening tool for behavioural and emotional problems
[SHACK-S] Devereux Early Childhood Assessment for Preschoolers, Second Edition (DECA-P2) [Experiences and Support Needs of Siblings of Critically Ill Children] | 1-, 3-, and 6-month post-PICU discharge
  Measures of social and emotional health and resilience, and screening for behavioural concerns (For siblings ages 4-5 years old)
[SHACK-S] KidCOPE [Experiences and Support Needs of Siblings of Critically Ill Children] | 1-, 3-, and 6-month post-PICU discharge
  Measure of cogntive and behavioural coping in children and adolescents (For siblings ages 6-18 years old)
[SHACK-S] Semi-structured interview [Experiences and Support Needs of Siblings of Critically Ill Children] | 3- and 6-month post-PICU discharge
  To understand experiences and support needs of siblings of critically ill children

SECONDARY OUTCOMES:
[HOPE] PedsQL 1.0 Infant Scales [Overall Family Health] | Baseline, Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measure generic health-related quality of life in infants (Only for study participants aged below 2 years old)
[HOPE] PedsQL 4.0 Short Form 15 (SF15) [Overall Family Health] | Baseline, Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measure generic health-related quality of life in children (Only for study participants aged 2 - 16 years old)
[HOPE] PedsQL 3.0 Cognitive Functioning Scales [Overall Family Health] | Baseline, Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measures cognitive functioning in paediatric patients (Only for study participants aged 2 - 16 years old)
[HOPE] PedsQL 2.0 Family Impact Module [Overall Family Health] | Baseline, Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Measures the impact of pediatric chronic health conditions on parents and the family
[HOPE] Patient Health Questionnaire-4 (PHQ-4) [Overall Family Health] | PICU discharge, Hospital Discharge (up to 18 months post-PICU discharge), 6-, 12- and 18-month post-PICU discharge
  Brief screener for depression and anxiety (in parent)
[HOPE] PTSD Checklist for DSM-5 [Overall Family Health] | 6-, 12- and 18-month post-PICU discharge
  Parent self-report measure of DSM-5 symptoms of PTSD

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Lee Jan Hau, MBBS, MRCPCH, MCI, Principal Investigator — KK Women's and Children's Hospital
Locations (2):
- Singapore (2):
  - National University Singapore, Singapore, Singapore
  - KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No